CLINICAL TRIAL: NCT07140549
Title: Survey of Patients Who Underwent Testicular Tissue Cryopreservation for Fertility Preservation Prior to Gonadotoxic Therapy in Childhood or Peripuberty
Brief Title: Survey of Patients Who Received Fertility Preservation Counseling and Underwent Testicular Tissue Cryopreservation Prior to Gonadotoxic Treatment During Childhood or Peripuberty
Acronym: QUALIFERT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023/14JUI/263
Record Dates: First submitted 2025-07-10; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-07

CONDITIONS: Satisfaction Survey; Fertility Perservation
Keywords: fertility preservation; boys; gonadotoxic treatment; male infertility; testicular tissue biopsy; spermatogonial stem cell; cryopreservation; long-term follow-up; survey
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who underwent gonadotoxic treatment for oncological or benign disease (Experimental): This survey study aims to assess the long-term outcomes and patient satisfaction of men who underwent a fertility preservation procedure i.e., a testicular biopsy with cryopreservation of immature testicular tissue, during prepuberty or peripuberty at the Cliniques Universitaires Saint Luc (CUSL) since the start of the fertility preservation program in 2005. Participants will be asked about their current reproductive health status, their experience with the fertility preservation process, and their overall satisfaction with the care they received.
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — A monocentric experimental study conducted as a survey, including patients enrolled in our fertility preservation program between May 2005 and May 2020.
  Participants were asked about their current reproductive health status, their experience with the fertility preservation process, and their overall satisfaction with the care they received.

SUMMARY:
Chemotherapy and radiotherapy can lead to spermatogonial stem cell depletion in pre- and peripubertal boys, potentially resulting in infertility during adulthood A testicular biopsy is considered a safe procedure performed in children prior to gonadotoxic treatment as part of a fertility preservation strategy. At the time of the procedure, parental involvement is essential-both in their role as legal guardians and due to the limited cognitive capacity of young boys to fully comprehend fertility preservation counseling.

Long-term follow-up is necessary to evaluate the impact on fertility outcomes, psychological well-being, and overall satisfaction. The aim of this survey is to assess the perceived impact of fertility preservation counseling and the physical and emotional effects of undergoing testicular biopsy in this population, with the goal of identifying opportunities to improve patient experience and clinical care for future patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have participated in the fertility preservation program aged 18 years old and above

Exclusion Criteria:

* Deceased patients. Patients undergoing treatment for disease relapse. Patients suffering from a documented mental disorder.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The impact on quality of life of fertility preservation during childhood or adolescence. | From the start of the program in may 2005 and the last patient enrolled in may 2020
  Assessment will be conducted by means of a confidential survey in > 18 yo patients who have undergone in their childhood a fertility preservation.
  The number of patients who are eligible for the follow-up survey (n = 64) within the fertility preservation program of the CUSL is important compared to the overall number of boys who have participated in such a FP programme worldwide (n=1033) in 2023.
  Recipients' satisfaction level will be evaluated by both general and specific scores. The general satisfaction score is calculated by combining the responses to questions rating specifically recipients' satisfaction on specific items using a 5 elements Likert scale (Very Dissatisfied to Very Satisfied) and responses to closed questions which inquire participants' global satisfaction on specific subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Wyns, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided